CLINICAL TRIAL: NCT02959008
Title: Continous Assessment of Cerebral Autoregulation With Near-infrared Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yu Liyun (Other)
Responsible Party: Sponsor-Investigator, Yu Liyun, Principal Investigator, Beijing Electric Power Hospital
Organization: Beijing Electric Power Hospital (Other)
Other Study IDs: 111
Record Dates: First submitted 2016-11-05; First posted 2016-11-08 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Cerebral Blood Flow; Cerebral Perfusion Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- normal: Human without hypertension, diabetes, anemia, liver disease and kidney disease. The group will measure TOI and BP.
  Interventions: Device: measure TOI and BP
- hypertension: Human only have hypertension, without diabetes, anemia, liver disease and kidney disease.
  Hypertension group will measure TOI and BP.
  Interventions: Device: measure TOI and BP

INTERVENTIONS:
Device: measure TOI and BP — Both groups measure TOI and BP.

SUMMARY:
Cerebral autoregulation can be explained by a tight coupling between oxygen supply and demand of the brain, and is essential to maintain a constant cerebral blood flow (CBF) in the context of changes in cerebral perfusion pressure. In this study, investigators use Near-infrared spectroscopy (NIRS) to monitor cerebral autoregulation.

DETAILED DESCRIPTION:
Near-infrared spectroscopy (NIRS) is a noninvasive technology that real-time monitors cerebral tissue oxygenation index (TOI). Investigators use Near-infrared spectroscopy (NIRS) to monitor cerebral autoregulation of hypertensive participants and non-hypertensive participants.

ELIGIBILITY:
Inclusion Criteria:

* health people, or people with hypertension

Exclusion Criteria:

* diabetes, anemia, liver disease, kidney disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. adult
  2. health people
  3. people with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
range of cerebral autoregulation | 30min

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohong Wu, Principal Investigator — Beijing Electric Power Hospital

IPD SHARING:
Plan to Share IPD: No